CLINICAL TRIAL: NCT02079727
Title: A Multicentre, Comparative, Randomised, Double-blind, Double-dummy Clinical Trial on the Efficacy and Safety of Condrosulf Versus Celebrex and Versus a Placebo in the Treatment of Knee Osteoarthritis
Brief Title: Condrosulf vs Celebrex vs Placebo in the Treatment of Knee OA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12EU/Ct06; 2013-001619-62 (EudraCT Number)
Record Dates: First submitted 2014-02-28; First posted 2014-03-06 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Knee Osteoarthritis
Keywords: Condrosulf; Chondroitin sulfate; Celebrex; Knee OA; Knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Chondroitin Sulfates; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Condrosulf (Chondroitin 4&6 sulfate) (Experimental): 1 tablet of Condrosulf 800 mg and 1 capsule of placebo of Celebrex once a day for 182 days
  Interventions: Drug: chondroitin sulfate
- Placebo (PBO) 800 mg tablet and Placebo (PBO) 200 mg capsule (Placebo Comparator): 1 tablet of PBO of Condrosulf and 1 capsule of PBO of Celebrex, once a day for 182 days
  Interventions: Drug: placebo
- Celebrex 200 mg capsule (Active Comparator): 1 capsule of 200 mg of Celebrex and 1 tablet of 800 mg placebo of Condrosulf once a day for 182 days
  Interventions: Drug: celecoxib

INTERVENTIONS:
Drug: chondroitin sulfate
  Other Names: Condrosulf
  Arms: Condrosulf (Chondroitin 4&6 sulfate)
Drug: celecoxib
  Other Names: Celebrex
  Arms: Celebrex 200 mg capsule
Drug: placebo
  Other Names: placebo for chondroitin sulfate and placebo for celecoxib
  Arms: Placebo (PBO) 800 mg tablet and Placebo (PBO) 200 mg capsule

SUMMARY:
The purpose of this study is to confirm the efficacy and safety of 800 mg Chondroitin 4&6 sulfate (Condrosulf) vs placebo once a day for 6 months in the symptomatic treatment of knee osteoarthritis. A third group, Celecoxib 200 mg (Celebrex) once a day, will be used as active comparator.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients of either sex, aged ≥50 years
* Patients affected by primary knee osteoarthritis of the medial or lateral femoro-tibial compartment
* Diagnosis according to the American College of Rheumatology (ACR) criteria
* Kellgren & Lawrence grade I-III
* Knee osteoarthritis evolving for more than 6 months
* Patients suffering from regular pain and functional disorders from at least 3 months
* Accomplishing a score ≥ 7 of Lequesne's index for the knee osteoarthritis
* Assessing pain on Huskisson's VAS ≥ 50 mm
* With radiography dated less than six months showing a remaining articular joint space
* Without such an axial disorder to justify an osteotomy
* Women taking contraceptive measures if not in menopause
* Women having negative pregnancy test
* Patients able to understand and follow the study protocol
* Patients who have signed the written informed consent for their participation in the clinical trial

Exclusion Criteria:

* With a history of heart attack, ischemic heart disease or cerebrovascular disease (including transient ischemic attacks)
* Having or have had peripheral arterial disease or past surgery orf peripheral arteries
* With a history or currently significat coagulation defect or/and blood dyscrasia
* With high risk of cardiovascular events
* With any acute or chronic infections requiring antimicrobial therapy or serious viral (e.g., hepatitis, HIV positivity) or fungal infections
* With a history of recurrent gastrointestinal ulceration or active inflammatory bowel diseases (e.g., Crohn's disease or ulcerative colitis)
* Having been diagnosed as having or have been treated for oesophageal, gastric, pyloric channel, or duodenal ulceration within 30 days prior to receiving the first dose of study medication
* Having severe liver or kidney disease
* With allergy to Celebrex or any of the other ingredients of Celebrex
* Having had an allergic reaction to sulphonamides
* Having had, as a result of intake of acetylsalicylic acid or other NSAIDs, asthma, nose polyps, severe nose congestion, or an allergic reaction such as itchy skin rash, swelling of the face, lips, tongue or throat, breathing difficulties or wheezing
* Presenting lactose intolerance
* Mild or not symptomatic knee osteoarthritis : < 7 of Lequesne's index,
* Pain on Huskisson's VAS (Visual Analogic Scale) < 50 mm
* Predominantly femoro-patellar osteoarthritis
* Destructive osteoarthritis of the knee justifying a surgery in the following 6 months
* Osteoarthritis with hydrarthrosis requiring a puncture or an infiltration
* Important genu varum or valgus >8° (physiological angle including)
* Kellgren & Lawrence grade IV
* Knee joint surgery in the last 3 months (e.g. chondroscopy, arthroscopy)
* Viscosupplementation, tidal lavage in the last 6 months
* Arthritis and metabolic arthropathies, Paget's illness
* Having consumed: basic treatment of arthritis with SYSADOA, symptomatic slow acting drugs for osteoarthrithis (chondroitin sulphates, glucosamine sulphates, diacerhein, hyaluronic acid and food supplement for joint care) in the last 3 months; treatment with corticoids, by any administration route during the last month; any medication having an influence on pain:
* NSAIDs (nonsteroidal anti-inflammatory drugs) in the 5 days preceding the inclusion (wash-out period considering 5 half-lives of the drug)
* hypnotics, muscle relaxants, anxiolytics, if the intake has started less than 8 days before inclusion
* paracetamol in the 10 hours preceding the inclusion
* Foreseen physiotherapy, re-education, alternative medicine (mesotherapy, acupuncture) in the next six months (study period)
* Presenting psychiatric illness hindering the protocol complaince, alcoholism, ongoing or < 1 year drug dependency
* Pregnant or likely to become it during clinical trial or lactating
* Women having positive pregnancy test
* Having participated in other clinical trials in the month preceding the clinical trial.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 604 (Actual)
Dates: Start 2014-06-12 (Actual); Primary Completion 2015-10-19 (Actual); Study Completion 2016-06-16 (Actual)

PRIMARY OUTCOMES:
Lequesne's Index | Day 1 and Day 182
  Decrease in the scores of the Lequesne's Index from Day 1 to Day 182.
Pain (VAS in mm) | Day 1 and Day 182
  Decrease in the VAS (pain in mm) from Day 1 to Day 182

SECONDARY OUTCOMES:
Lequesne's Index | Day 1, 30, 90 and 182
  Evolution from Day 1 to Day 30, Day 90 and Day 182
Pain (VAS in mm) | Day 1, 30, 91 and 182
  Evolution of the pain on VAS (in mm) from Day 1 to Day 30, Day 91 and Day 182
MCII (minimal clinically important improvement) | Day 1, 30, 91 and 182
PASS (patient acceptable symptom state) | Day 1, 30, 91 and 182
Consumption of Paracetamol | Day 1, 30, 91 and 182
Global efficacy assessment | At Day 30, 91 and 182
  Global efficacy assessed by the patient and the Investigator by means of a semi-quantitative verbal scale.
Number of adverse events related to the treatments | At Day 30, 91 and 182
Number of drop-outs due to AE (adverse event) related to the treatment | At Day 30, 91 and 182

OTHER OUTCOMES:
Treatment compliance | Day 1, 30, 91 and 182

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves Reginster, Prof. MD PhD, Principal Investigator — Unité d'Exploration du Métabolisme Osseux, CHU Centre ville, Polycliniques Universitaires L-Brull, Liège, Belgium
Locations (16):
- Unité d'exploration du metabolism osseux, CHU, Polyclinique universitaires L-Brull, Liège, Liege, Belgium
- Czechia (6):
  - Ortopedicka Ambulance, Brno
  - Interni a revmatologicka ordinace, Břeclav
  - Vesalion s.r.o., Ostrava
  - Revmatologicky ustav, Prague
  - Thomayerova nemocnice - Revmatologicke a rehabilitacne oddeleni, Praha - Krc
  - Medical Plus, Uherské Hradiště
- Azienda Osp. Univ. Di Careggi, Florence, Italy
- Poland (5):
  - Klinika Zdrowej Kosci, Lodz
  - Lubelskie Centrum Diagnostyczne, Świdnik
  - SOLB, Ul. Jana III Sobieskiego
  - Medica Pro Familia, Warsaw
  - Zdrowie Osteo-Medic, Wiejska
- Switzerland (3):
  - Bethesda-Spital, Basel
  - HFR Fribourg - Hôpital Cantonal, Fribourg
  - Universitätsspital Zürich, Rheumaklinik, Zurich